CLINICAL TRIAL: NCT01429766
Title: A Prospective Study of Variation in Breath Holding Times at Various Phases of Respiration During the Course of Radiotherapy Including the Effect of Respiratory Training in Lung Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Anusheel Munshi, Associate Professor, Tata Memorial Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 747
Record Dates: First submitted 2011-08-25; First posted 2011-09-07 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Small Cell Lung Cancer; Non Small Cell Lung Cancer
Keywords: Breath holding times; Phases of respiration; Radiotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Respiratory Training — All patients shall be sent for respiratory training to the physiotherapy department. Patients shall be counseled about respiratory training by trained staff in their own vernacular. Whenever possible, patients shall be provided one "Spiroball" device and taught how to use the device. In addition/alternatively patients will be taught to do pranayam(breath exercises). Patients provided with spiroball shall be instructed to use the spiroball by the prescribed technique. The following visit schedule shall be observed
  1. st visit Within one day of the date of simulation
  2. nd visit Date of Radiotherapy start Subsequently 2 visits per week during radiotherapy course shall be conducted (Tuesdays, Thursdays)

SUMMARY:
100 suitable patients of lung cancer shall be taken into the study over a period of 2 years. As per the existing treatment protocol in our department, all patients suitable shall undergo a routine Pulmonary function testing (PFT). Subsequently, recording of the breath hold shall be done at the following times

1. At time of simulation
2. At the time of first fraction of radiotherapy
3. At mid radiotherapy
4. At radiotherapy conclusion After the recording at a), patients shall be asked to perform deep breathing exercises/spirometer ball exercise to see the effect of training on the breath holding times.

DETAILED DESCRIPTION:
100 suitable patients of lung cancer shall be taken into the study over a period of 2 years. As per the existing treatment protocol in our department, all patients suitable shall undergo a routine Pulmonary function testing (PFT). Subsequently, recording of the breath hold shall be done at the following times

1. At time of simulation
2. At the time of first fraction of radiotherapy
3. At mid radiotherapy
4. At radiotherapy conclusion After the recording at a), patients shall be asked to perform deep breathing exercises/spirometer ball exercise to see the effect of training on the breath holding times.

Respiratory training All patients shall be sent for respiratory training to the physiotherapy department. Patients shall be counseled about respiratory training by trained staff in their own vernacular. Whenever possible, patients shall be provided one "Spiroball" device and taught how to use the device. In addition/alternatively patients will be taught to do breath exercises. Patients provided with spiroball shall be instructed to use the spiroball by the prescribed technique. The following visit schedule shall be observed

1. st visit Within one day of the date of simulation
2. nd visit Date of Radiotherapy starting Subsequently 2 visits per week during radiotherapy course shall be conducted (Tuesdays, Thursdays) During all the above visits , respiratory training shall be reinforced and objective recording of the spirometer ball(whenever used) shall be recorded.(Inspiratory volume)

The breathing exercises shall continue through radiotherapy. At all the above times, recording shall be made of the breath holding times. In general at the start of each recording a nasal clip shall be placed and the patient shall be asked to close the mouth voluntarily. The closure of the mouth shall be done after nasal clip placement and then stopwatch for recording shall be started. The end time shall be the moment when the patient opens his mouth and starts breathing again. A one minute pause shall be kept between separate recordings.

1. Deep inspiratory breath hold(DIBH): A clip shall be placed on the nose. The patient shall be asked to take a deep breath from his mouth and then hold his breath.
2. Deep expiratory breath hold(DEBH): A clip shall be placed on the nose. The patient shall be asked to exhale maximally from the mouth and then hold his breath.
3. Normal mid ventilation breath hold(NVBH): A clip shall be placed on the nose. The patient shall be asked to hold breath in the middle of normal respiration.

Beam on/off times As mentioned before, all the patients shall be treated as per existing departmental protocol. However, as a planning component of the study, after the patients have been planned as per the routine protocol, the breath hold data in each phase shall be used to calculate the number of times the radiation beam would have to be needed if patients were treated with the above breath hold timings.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of Small cell and Non small cell lung cancer
2. Patients posted for 3DCRT or IMRT or IGRT

Exclusion Criteria:

1. Patients, who in view of their advanced disease and/or poor general condition would not be able to tolerate radical RT.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Breath holding time in various phases of the respiratory cycle | 2 years
  Breath holding time in deep inspiration, mid ventilation and end expiration

CONTACTS AND LOCATIONS:
Overall Officials: Anusheel Munshi, MD, Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

REFERENCES:
- See also: Web site of Tata Memorial Hospital — http://tmc.gov.in